CLINICAL TRIAL: NCT05253547
Title: Dietary Intervention Study on Food Based Dietary Guidelines for Sustainable and Healthy Lifestyles
Acronym: SuHeGuide
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College Dublin (Other)
Collaborators: Teagasc (Industry); University College Cork (Other); Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Aifric O'Sullivan, Lecturer/Assistant Professor, University College Dublin
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: LS-21-51-Davies-OSullivan
Record Dates: First submitted 2022-02-08; First posted 2022-02-23 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Dietary Habits; Healthy Diet; Healthy Nutrition; Personalized Nutrition
Keywords: Sustainable diets; Greenhouse gas emissions; Climate-friendly; Personalized nutrition
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Parallel randomized control trial
Who Masked: Participant
Masking Description: Single-blinded parallel study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy climate-friendly dietary guidelines (Experimental): Personalised healthy dietary recommendations aimed at reducing diet-related greenhouse gas emissions
  Interventions: Behavioral: Healthy climate-friendly dietary guidelines
- Healthy eating guidelines (Active Comparator): Personalised healthy dietary recommendations based on Ireland's Healthy Eating Guidelines
  Interventions: Behavioral: Healthy dietary guidelines

INTERVENTIONS:
Behavioral: Healthy climate-friendly dietary guidelines — Personalised climate-friendly healthy dietary recommendations
  Arms: Healthy climate-friendly dietary guidelines
Behavioral: Healthy dietary guidelines — Personalised healthy dietary recommendations
  Arms: Healthy eating guidelines

SUMMARY:
The aim of the study is to provide proof of the effectiveness, acceptability, healthfulness and nutritional adequacy of dietary guidelines to reduce greenhouse gas emissions. The study will compare the effect of dietary advice based on 1) healthy climate-friendly dietary guidelines (intervention group) or 2) standard healthy dietary guidelines (control) on greenhouse gas emissions associated with dietary intake over 12 weeks.

DETAILED DESCRIPTION:
A randomised, parallel controlled trial will recruit n=360 healthy adults (age 18-64) across three research centres. After successful screening and receiving informed consent, participants will be randomised into the intervention or the control group for the duration of the 12-week trial described in detail in the text and figure below. The intervention group will receive dietary advice based on climate friendly eating recommendations. The control group will receive dietary recommendations based on Healthy Ireland's Healthy Eating Guidelines and Food Pyramid (FSAI, 2019).

Prior to their first onsite visit, participants will be asked to complete a Health and Lifestyle questionnaire and dietary assessment. The dietary assessment will include

1. 3 online 24-hour recalls (2 non-consecutive weekdays and 1 weekend day) (via web-based dietary recall tool, Foodbook24)
2. a food frequency questionnaire (Foodbook24)

Baseline, Visit 1 (Week 0): We will collect blood and urine samples from participants and record anthropometric measurements. Participants will be asked to complete a Stage of Change questionnaire to assess their openness to a diet change. All participants will complete a Food Waste Questionnaire at baseline for later comparison at endpoint. At the end of Visit 1 participants will receive a personalised feedback report and advice from nutritionists based on their habitual diet.

Week 6: Participants will be asked to complete a second dietary assessment during week 6. 3 24-hour recalls and a food frequency questionnaire will be hosted on Foodbook24, a web-based dietary recall tool.

Week 11: Before attending endpoint onsite visit, participants will complete a final dietary assessment. The same assessment as Pre-baseline and Week 6 will be used.

Endpoint, Visit 2 (Week 12): At the end of 12 weeks, participants will be invited back for a follow-up assessment. Blood and urine samples and anthropometrics will be collected/recorded. Participants will complete the Stage of Change questionnaire and Food Waste questionnaire. A Tolerance questionnaire will be administered to see how willing participants would be to continue with their prescribed diet.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* Be a healthy adult between the ages of 18-64 years old
* Consume a diet associated with moderate-high greenhouse gas emissions
* Be in good general health

Exclusion Criteria:

* Are pregnant, lactating or planning to become pregnant
* Are following a medically prescribed diet
* Have a diagnosis of an acute or chronic medical condition that could interfere with the outcomes of the study. Such diagnoses include (but are not limited to) cardiovascular disease, diabetes mellitus, inflammatory bowel disease, cancers (within the last 5 years), etc.
* Are immunocompromised or have a suspected immunodeficiency
* Have excessive alcohol intake (>28 units per week)
* Have a known food allergy
* Regularly consume a single high-dose vitamin or mineral supplement
* Are participating in another research study
* Are unable to read, write or understand English.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 355 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Diet-related greenhouse gas emissions reported as kilograms of carbon dioxide equivalents per day | 12 weeks
  Participants will record their diet at baseline (habitual diet) and endpoint (intervention diet) using an online 24-hour recall method. Diet-related greenhouse gas emissions will be estimated using food, nutrient and food-related greenhouse gas emissions databases (measured as kilograms of carbon dioxide equivalents). The primary outcome measure is the change in diet-related greenhouse gas emissions (kgCO2-eq/day) as a result of the intervention diet.

SECONDARY OUTCOMES:
Calcium intake (milligrams per day) | 12 weeks
  Calcium intake will be calculated using dietary intake records (3x 24-hour recalls) at baseline and endpoint (intervention diet). The secondary outcome measure is the change in calcium intake (mg/day) as a result of the intervention diet.
Iron intake (milligrams per day) | 12 weeks
  Iron intake will be calculated from dietary intake records (3x 24-hour recalls) at baseline and endpoint (intervention diet). The secondary outcome measure is the change in iron intake (mg/day) as a result of the intervention diet.
Urinary iodine (micrograms per liter) | 12 weeks
  Participants will provide urine samples at baseline (Week 0) and endpoint (Week 12). Urinary iodine concentrations (ug/L) will be measured. The secondary outcome measure is the change in urinary iodine as a result of the intervention diet.
Serum vitamin D status (25(OH)D nanomole per liter) | 12 weeks
  Participants will provide blood samples at baseline (Week 0) and endpoint (Week 12). 25(OH)D will be measured (nmol/L) as a marker of vitamin D status. The secondary outcome measure is the change in vitamin D as a result of the intervention diet.
Serum lipids (milimoles per liter) | 12 weeks
  Participants will provide blood samples at baseline (Week 0) and endpoint (Week 12). Serum lipids, including total cholesterol, HDL cholesterol and triglycerides (mmol/L) will be measured. The secondary outcome measure is the change in lipid profile as a result of the intervention diet.
Fasting glucose (milimoles per liter) | 12 weeks
  Participants will provide blood samples at baseline (Week 0) and endpoint (Week 12). Fasting blood glucose will be measured (mmol/L). The secondary outcome measure is the change in fasting glucose as a result of the intervention diet.

CONTACTS AND LOCATIONS:
Overall Officials: Aifric O'Sullivan, PhD, Principal Investigator — University College Dublin
Locations (3):
- Ireland (2):
  - University College Cork, Cork
  - University College Dublin, Dublin
- Queen's University Belfast, Belfast, United Kingdom

IPD SHARING:
Plan to Share IPD: No
At the start of the study each participant will have a study code assigned to them. All of the data from the trials will be stored using these unique study codes. A file will be set up which will be stored in a location separate to the study data. This file will contain a list which will link each participants contact details to the corresponding ID code. All stored information will be encrypted and protected by a password that only the researcher and PI will know.

REFERENCES:
- [Derived] Davies KP, Gibney ER, Leonard UM, Lindberg L, Woodside JV, Kiely ME, Nugent AP, Arranz E, Conway MC, McCarthy SN, O'Sullivan AM. Sustainable diets reduce diet-related greenhouse gas emissions and improve diet quality: results from the MyPlanetDiet randomized controlled trial. Am J Clin Nutr. 2025 Oct;122(4):962-971. doi: 10.1016/j.ajcnut.2025.05.015. Epub 2025 Aug 26. PMID 41043876
- [Derived] Leonard UM, Davies KP, Lindberg L, Woodside JV, Nugent AP, O'Sullivan AM, Gibney ER, McCarthy SN, Arranz E, Kiely ME. Impact of sustainable diets on micronutrient intakes and status: outcomes of the MyPlanetDiet randomized controlled trial. Am J Clin Nutr. 2025 Nov;122(5):1275-1288. doi: 10.1016/j.ajcnut.2025.09.009. Epub 2025 Sep 8. PMID 40930463
- [Derived] Davies KP, Gibney ER, Leonard UM, Lindberg L, Woodside JV, Kiely ME, Nugent AP, Arranz E, Conway MC, McCarthy SN, O'Sullivan AM. Developing and testing personalised nutrition feedback for more sustainable healthy diets: the MyPlanetDiet randomised controlled trial protocol. Eur J Nutr. 2024 Oct;63(7):2681-2696. doi: 10.1007/s00394-024-03457-0. Epub 2024 Jul 6. PMID 38970665